CLINICAL TRIAL: NCT00329810
Title: A Prospective, Multicenter, Open-Label Study to Evaluate the Effectiveness and the Effect on Cognitive Function of a Treatment With Aripiprazole in a Board Range of Schizophrenic Patients
Brief Title: Effect on Cognitive Function of a Treatment With Aripiprazole
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN138-166
Record Dates: First submitted 2005-09-12; First posted 2006-05-25 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2012-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

ARMS (1):
- Switch (Experimental)
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Tablets, oral, 15 mg, once daily, 12 weeks.
  Other Names: Abilify

SUMMARY:
To evaluate the effectiveness of Aripiprazole after 12 weeks of therapy for Schizophrenic patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia
* score of 2-6 in the CGI-S scale at basline
* ambulatory or hospitalized subjects having symptoms which requires antipsychotic treatment

Exclusion Criteria:

* women of child bearing potential
* women pregnant or breast feeding
* patients with a score of 0,-1 or 7
* substance use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2005-03; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression scale at endpoint

SECONDARY OUTCOMES:
Change in Clinical Global Impression scale and cognition scales at endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Principal Investigator — Bristol-Myers Squibb

REFERENCES:
- [Derived] Bervoets C, Morrens M, Vansteelandt K, Kok F, de Patoul A, Halkin V, Pitsi D, Constant E, Peuskens J, Sabbe B. Effect of aripiprazole on verbal memory and fluency in schizophrenic patients : results from the ESCAPE study. CNS Drugs. 2012 Nov;26(11):975-82. doi: 10.1007/s40263-012-0003-4. PMID 23018547